CLINICAL TRIAL: NCT04754178
Title: Assessment of Skills and Behaviors in Children With Down Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal Investigator; PT; PhD, Universidad de Granada
Other Study IDs: DF0093UG
Record Dates: First submitted 2021-02-11; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Down syndrome: Down syndrome patients and their parents
- Control group: Healthy children and their parents

SUMMARY:
Parents of children with Down Syndrome can help in describing children's abilities and behavior. Most of the studies evaluating parents of children with Down Syndrome and other intellectual disabilities have focused on parental stress and coping; Additionally, most research has evaluated the perspectives of mothers rather than fathers. For this reason, in this study we aims to evaluate skills and behaviors in children with Down syndrome through the perception of parents.

ELIGIBILITY:
Inclusion Criteria:

* Down syndrome childrens
* Age between 0 and 3 years

Exclusion Criteria:

* Other physical or functional impairment that limits the performance of evaluation

Ages: 0 Years to 3 Years | Sex: All
Age Groups: Child
Study Population: Patients with Down Syndrome
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
Early Motor Questionnaire | Baseline
  The EMQ is designed as a fast and easy to complete motor questionnaire, and is organized into 3 sections: Gross motor skills, fine motor skills, and perception-action integration skills. The EMQ is not a standardized assessment, but can be used in research settings, serve as a motor screener, or as complement to standardized measures of early motor development.
Montreal's children's Hospital Feeding Scale | Baseline
  The Montreal Children's Hospital Feeding Scale (MCHFS) is a quick and reliable measure of feeding problems for clinical settings, but there is little examination of its relationship to commonly used research measures of parental feeding practice, child eating behaviour and observations of parent-infant interaction at mealtimes.
Feeding Hándicap Índex Children | Baseline
  y the Feeding Handicap Index (FHI), [20] was developed and standardized on typically developing children, children with CP, Autism spectrum disorder in the age range of 2-10 years and Intellectual disability. FHI has 38 items related to statements related to physical (21), emotional (12) and functional (5) aspects of feeding and swallowing abilities. It has a 3 point rating scale (0, 1 & 2) where "0" indicates the individual "Never has this problem", "1" indicates "Sometimes has this problem" and "3" indicates "Always has this problem"
Parent Perceptions of Physical Activity Scale | Baseline
  Evaluate the Parent Perceptions of Physical Activity in Families of Toddlers With Neurodevelopmental Disorders
Bayley Scales of Infant and Toddler Development | Baseline
  is an individually administered scale that assesses five key developmental domains in children between 1-42 months of age: cognition, language (receptive and expressive communication), motor (gross and fine), social-emotional and adaptive behavior. The first three are assessed through direct observation of the child in test situations, while the last two are assessed through questionnaires to be completed by the main caregiver.
Early Clinical Assessment of Balance | Baseline
  The Early Clinical Assessment of Balance (ECAB) is a measure of postural stability for children.
Infant Positioning Assessment Tool | Baseline
  The Infant Position AssessmentTool (IPAT) is a six-item tool with cumulative scores ranging from 0 to 12. It was developed as a teaching tool to standardize developmentally supportive positioning practices in the NICU and provides a method for evaluation of those positioning practices.
Asymmetry | Baseline
  Asymmetry was evaluated with photography
COMFORT behaviour scale | Baseline
  The COMFORT behaviour scale (COMFORT-B scale) is widely used in paediatric intensive care units to assess young children's pain and distress.
Segmental Assessment of Trunk Control | Baseline
  The SATCo i,ii is a validated outcome measure that identifies at which head/trunk segment Targeted Training should commence. The SATCo determines the topmost (most cephalo) segment at which control of the upright posture is poor or not demonstrated i.e. is currently being learned for each of static, active and reactive control.

SECONDARY OUTCOMES:
EuroQol-5D | Baseline
  The perception of the level of health and the quality of life were evaluated with the questionnaire European Quality of
  Life-5 Dimensions (EQ-5D). It is composed of 2 parts in which health status is assessed:
  * Descriptive system: It consists on 5 dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Patients classify their health status in 3 severity levels: having no problems, having some or moderate problems, being unable to do/having extreme problems.
  * Visual Analog Scale, by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status)
Hospital Anxiety and Depression Scale | Baseline
  Anxiety and depression will be assessed with the Hospital Anxiety and Depression Scale (HADS) . This scale is composed of 14 items divided into two subscales, 7 items of anxiety and 7 items of depression, involving higher values worse psycho-emotional state
Zarit Burden Interview | Baseline
  The Zarit Burden Interview, is a popular caregiver self-report measure used by many aging agencies. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always).
International physical activity questionnaire | Baseline
  The International Physical Activity Questionnaire (IPAQ) was developed to measure health-related physical activity (PA) in populations.
Charlson comorbidity index | Baseline
  Charlson Comorbidity Index predicts the ten-year mortality for a patient who may have a range of comorbid conditions
Brief Infant Sleep Questionnaire | Baseline
  The Brief Infant Sleep Questionnaire (BISQ) is used to assess sleep patterns, parent perception, and sleep-related behaviors in young children (0-36 months). The BISQ has been validated against actigraphy, daily logs, and has high sensitivity in documenting expected developmental trends in sleep

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Healthy Sciences, Granada, Spain

IPD SHARING:
Plan to Share IPD: No